CLINICAL TRIAL: NCT01078597
Title: A Study on the Prevalence of the Modified Citrullinated Vimentin Anti-body (Anti-MCV) in an Irish Rheumatoid Arthritis (RA) Population and to Assess the Impact of Anti-MCV and the Anti-cyclic-citrullinated Peptide Antibody (Anti-CCP) Status on the Management of Irish Patients With Early RA
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: JSS Medical Research Inc. (Industry); Clinical Trial End-Point (CTEP) Ltd (Unknown)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P11-983
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
Keywords: anti-MCV; anti-CCP; Biomarkers; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — There are no biospecimens specifically retained for the purposes of the study. Routine blood samples may be retained as per routine practice of the participating centre.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with early Rheumatoid Arthritis: Patients , aged 18 years or over, diagnosed with Rheumatoid Arthritis, with evidence of disease activity within the last year.

SUMMARY:
A key challenge in the management of patients with Rheumatoid Arthritis (RA) is the early identification of patients that are at risk of developing a severe and destructive disease. A better understanding of prognostic factors such as anti-CCP and anti-MCV biomarkers, is needed in order to better identify patients with early Rheumatoid Arthritis that are at risk of developing aggressive diseases. At the present time the prevalence of one such biomarker, namely anti-MCV, is unknown in an Irish Rheumatoid Arthritis population. This study will establish the prevalence of anti-MCV in such a population.

A second challenge in the management of Rheumatoid Arthritis patients is the determination of the best treatment strategy tailored to individual patient's needs. In routine practice, treatment approaches are based on the patient history and the availability of clinical parameters, such as a positive anti-CCP status, which is associated with worst prognostics. At the present time, the impact of a positive anti-CCP status on patients' management has not been formally studied in Ireland The proposed study will provide data on the prevalence of anti-MCV in an Irish RA population and the use of anti-CCP and other clinical parameters currently used in routine care. In addition, the present study will evaluate the impact of the known anti-CCP status on patients' management. Associations between the anti-CCP and anti-MCV status and clinical outcome measures will be assessed.

The results from the present study will have significant implications not only for the individual patient but also from the societal perspective, since it will enhance the overall understanding and applications of different treatment approaches based on individual patients' profile.

DETAILED DESCRIPTION:
Results from clinical studies suggest that approximately 73% of patients with Rheumatoid Arthritis present evidences of erosions within 2 years of the diagnosis. Early interventions with Disease Modifying Anti-Rheumatic Drug (DMARD) therapies have been shown to reduce the progression of the disease. Significant differences in mean Sharp scores were observed two years after the initiation of such treatment regimens. These data support the existence of a "therapeutic window", during which the rheumatoid process should be stopped or retarded in order to prevent further articular damages. Importantly, these observations constituted the premise of subsequent researches aiming at evaluating the benefits of TNF inhibitors in patients with early and aggressive rheumatoid arthritis.

The detection of soluble biomarkers indicates the occurrence of active changes in the underlying disease processes. Recently, the OMERACT group has undertaken the task of developing validation criteria for biomarkers. Validated biomarkers will be considered reliable surrogate measures of radiological endpoints. C Reactive Protein (CRP) has recently been validated using those newly developed criteria (ACR 2006). Noteworthy, the association of CRP with damage endpoints appears to vary based on the use of different anti-rheumatic medications. Other soluble biomarkers, which are being used in routine care, will be soon evaluated against those same criteria.

Several other biomarkers of interest, including serum MMP-3, urinary CTX-II, serum OPG/RANKL, serum CEC, and the CPII/C2C ratio, are being extensively evaluated in various clinical studies. A recent study evaluated antibodies against modified citrullinated vimentin (anti-MCV).

Predictors/prognostic markers indicate the presence of a change in the underlying disease processes. However, their value is mainly related to their reliability at predicting future changes, such as the clinical onset of the disease, the severity of the disease or associated complications. In this respect, they are early indicators of future events.

Rheumatoid factors (RFs) are autoantibodies directed towards the Fc portions of IgG. RFs are found in multiple immunoglobulin isotypes (IgE, IgM, IgA and IgG), however, IgM is the isotype that is preferentially measured in clinical assays. RFs have long been associated with the development and the severity of RA. The sensitivity and the specificity of RF in the diagnosis of RA have been shown to be close to 60% and 79%, respectively. This is rather low comparatively to other prognostic markers. This is mainly because RF is also detected in normal healthy individuals as well as in various infections and other rheumatological illnesses. As a result, its individual diagnostic value appears to be unsatisfactory. This may be an issue in patients with early and undifferentiated arthritis. In this regard, IgM RFs has been shown to be positive in 19.3% of RA patients prior to the onset of their symptoms.

Antibodies targeting determinants resulting from the deamination of peptidylarginine to peptidyl citrulline residues have recently received a great deal of attention. These include antibodies directed against cyclic citrullinated peptide (anti-CCP) and antibodies targeting in vivo citrullinated proteins, such as anti-keratin antibodies, antiperinuclear factor, anti-citrullinated (pro)filaggrin and anti-Sa/citrullinated vimentin. The prognostic and predictive values of anti-CCP antibodies have been extensively reviewed elsewhere. These results indicate that anti-CCP antibodies are highly predictive of the future development of RA in both healthy individuals and patients with undifferentiated arthritis. A more recent study evaluated the sensitivity, specificity, and prognostic value of determination of levels of anti-MCV as compared with anti-CCP in an inception cohort of patients with early RA The findings showed that analysis of anti-MCV yields greater sensitivity and unchanged specificity as compared with analysis of anti-CCP. And also appears to perform better than anti-CCP in identifying poor radiographic prognosis in patients with early RA.

These observations suggest that different antibodies targeted against citrullinated agents may differ in their ability to predict poor outcomes. Collectively, these observations indicate that the predictive values of various predictors may be enhanced when combined with other predictors/prognostic markers of the disease.

Primary Objectives

* To describe the prevalence of anti-MCV in an Irish RA population
* To assess the association of anti-MCV with RF and anti-CCP in this population.
* To assess the impact of known anti-CCP status (positive or negative) and anti-MCV on clinical decision-making and the management of patients recently diagnosed with RA.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient was diagnosed with Rheumatoid Arthritis with evidence of disease activity within the past year.
* Patient has known anti-CCP status (positive or negative).
* Patient has agreed to participate in the study by signing an informed consent.
* Patient will be available for a period of follow-up of 12 months, from the time of enrollment in the study
* Patient is fluent in the English language

Exclusion Criteria:

* Patient's anti-CCP status (positive or negative) has not been determined.
* Patient with any other rheumatological disorder such as mixed connective tissue disease, psoriatic arthritis, ankylosing spondylitis, scleroderma and crystal induced arthropathies. Osteoarthritis is not an exclusion criterion.
* Patient with any condition that would prevent participation in the study and completion of the study procedures, including language limitation.
* Patient is not willing to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis attending specialist rheumatology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Anti-Cyclic Citrullinated Protein blood test results | Baseline (Week 0), 6 months, 12 months
Anti-Modified Citrullinated Vimentin blood test result | Baseline Visit (Week 0)
Rheumatoid Factor blood test result | Baseline (Week 0), 6 months, 12 months
Investigator Questionnaire assessing the impact (if any) of biomarker status on the management of the patient | Baseline (Week 0), 6 months, 12 months

SECONDARY OUTCOMES:
C- Reactive Protein (CRP) & Erythrocyte Sedimentation Rate (ESR) blood test results | Baseline (Week 0), 6 months, 12months
Swollen Joint Count | Baseline (Week 0), 6 months, 12 months
Tender Joint Count | Baseline (Week 0), 6 months, 12 months
Disease Activity Score (DAS)-28 | Baseline (Week 0), 6 months, 12 months
Health Assessment Questionnaire Disability Index (HAQ-DI) | Baseline (Week 0), 6 months, 12 months
Visual Analogue Scale-Disease Activity (VAS-DA) | Baseline (Week 0), 6 months, 12 months
Visual Analogue Scale - Pain (VAS-Pain) | Baseline (Week 0), 6 months, 12 months
Visual Analogue Scale - General Health (VAS-GH) | Baseline (Week 0), 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Mc Carthy, Principal Investigator — Mater Misercordiae Hospital, Dublin
Locations (4):
- Ireland (4):
  - Site Reference ID/Investigator# 49402, Cork
  - Site Reference ID/Investigator# 49403, Cork
  - Site Reference ID/Investigator# 22307, Dublin
  - Site Reference ID/Investigator# 72114, Dublin

REFERENCES:
- See also: Related Info — http://rxabbvie.com